CLINICAL TRIAL: NCT02854683
Title: Reducing Orthostatic Intolerance With Oral Rehydration in Patients With Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Brief Title: Reducing Orthostatic Intolerance With Oral Rehydration in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: New York Medical College (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: L-11-531-101; 1R21NS094644-01 (NIH)
Record Dates: First submitted 2016-07-29; First posted 2016-08-03 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Chronic Fatigue Syndrome; Myalgic Encephalomyelitis; Systemic Exertion Intolerance Disease (SEID); Postural Tachycardia Syndrome (POTS); Neurally Mediated Syncope (NMS)
Keywords: Chronic Fatigue Syndrome (CFS); Myalgic Encephalomyelitis (ME); Postural Tachycardia Syndrome (POTS); Neurally Mediated Syncope (NMS); Systemic Exertion Intolerance Disease (SEID); Orthostatic Intolerance (OI); Oral Rehydration Solution (ORS); Lower Body Negative Pressure (LBNP)
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Postural Orthostatic Tachycardia Syndrome; Syncope, Vasovagal; Orthostatic Intolerance; Osteoarthritis | interventions — Saline Solution; World Health Organization oral rehydration solution; ORALIT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal Saline (Experimental): Subjects will receive 1 liter of intravenous normal saline over 1 hour and on an alternate day Subjects will drink ORS solution 1 liter total by mouth over 20 minutes.
  Interventions: Drug: Normal Saline
- Oral rehydration solution (Experimental): Subjects will receive 1 liter of intravenous normal saline over 1 hour and on an alternate day Subjects will drink ORS solution 1 liter total by mouth over 20 minutes.
  Interventions: Dietary Supplement: Oral Rehydration Solution

INTERVENTIONS:
Drug: Normal Saline — 1 liter of intravenous saline will be delivered over 1 hour
  Other Names: NSS
  Arms: Normal Saline
Dietary Supplement: Oral Rehydration Solution — 1 liter of ORS solution given by mouth
  Other Names: ORS
  Arms: Oral rehydration solution

SUMMARY:
We and others have shown that many younger patients with Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) have orthostatic intolerance (OI), i.e., they can't tolerate prolonged standing. OI in ME/CFS is often accompanied by either postural tachycardia syndrome (POTS) in which standing results in an excessive heart rate, and neurally mediated hypotension (NMH) in which standing causes a fall in blood pressure and fainting. Intravenous fluids can alleviate these symptoms, but is difficult to administer; oral fluids fail to provide the same benefit. We would therefore like to test the effectiveness of an oral rehydration solution (ORS, W.H.O. formula) making use of co-transport of glucose and sodium, to reverse these symptoms in ME/CFS subjects with POTS or NMS, and will compare these results with healthy control subjects.

DETAILED DESCRIPTION:
We and others have shown that a majority of younger patients with Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) have orthostatic intolerance (OI), the inability to tolerate orthostatic stress such as prolonged standing. OI in ME/CFS comprises postural tachycardia syndrome (POTS) in which symptoms occur along with excessive upright heart rate, and neurally mediated hypotension (NMH) in which symptoms occur along with an upright fall in blood pressure. The causes of OI are diverse but are clearly initiated by postural contraction of central blood volume (BV) by gravitational translocation of 500-800 mL of blood from the upper to the lower body. Intravenous central BV expansion with isotonic saline is commonly and effectively used to reduce OI regardless of etiology, but has complications if used long term. Usual forms of oral hydration fail to provide similar benefit. Interestingly, a specific isotonic oral rehydration solution (ORS W.H.O. formula), making use of co-transport of glucose and sodium, has been shown to efficiently rehydrate cholera patients suggesting an ability to increase central BV rivaling intravenous fluids. Since the circulatory effects of saline or ORS BV expansion are incompletely understood, we propose to study the neurovascular physiology of fluid loading during orthostatic stress in ME/CFS patients with POTS or NMH, comparing results with healthy control subjects. We hypothesize that equal volumes of ORS is not inferior and may be superior to intravenous saline infusion in increasing intravascular and interstitial fluid volume and improving orthostatic tolerance. Using noninvasive measurements of heart rate and blood pressure by Finapres and oscillometry, cardiac output and peripheral arterial resistance by inert gas rebreathing, cerebral blood flow velocity by transcranial Doppler ultrasound, and regional fluid shifts by impedance and venous occlusion plethysmography, we have acquired preliminary data in ME/CFS patients with OI demonstrating superior restoration of orthostatic tolerance with ORS. We will recruit patients aged 15-29 years who have confirmed ME/CFS with OI, including 15 with NMH and 15 with POTS, and compare them to 15 healthy volunteer subjects. In Specific Aim 1 we will measure BV by Daxor iodinated albumin technique before orthostatic stress imposed by step-wise lower body negative pressure (LBNP) to measure the threshold for OI. Relative changes in BV using serial hematocrits in OI patients will be compared to data from control subjects similarly tested. In Specific Aim 2, all subjects will be randomized to receive saline or ORS in a cross over study. On one day, total BV and neurovascular properties will be measured in patients and control subjects before and 1 hour after completing one liter administration of intravenous normal saline infusion or ORS. On another day (separated by 1 week), we will repeat measurements using the other hydration route. We will perform LBNP on each day following saline or ORS to determine whether orthostatic intolerance and circulatory physiology are improved similarly with equivolumic IV saline or ORS hydration.

ELIGIBILITY:
Inclusion Criteria:

* Both female and male participants are being studies
* Ages 15-29
* All subjects must fulfill criteria for Myalgic Encephalomyelitis (ME)/Chronic Fatigue Syndrome (CFS) and include 15 with Neurally Mediated Syncope (NMS) and 15 with Postural Tachycardia Syndrome (POTS).
* ME/CFS patients with NMS will be cases with episodic symptoms of Orthostatic Intolerance (OI) associated with 3 or more episodes of abrupt loss of consciousness and postural tone within the last year (simple faint)
* ME/CFS patients with POTS will have chronic day to day symptoms of OI for at least 3 months. POTS will be confirmed by duplication of these symptoms per tilt table test
* Healthy volunteers will be included and free from any disease

Exclusion Criteria:

* all subjects will have normal physical exam and be free of all systemic disease
* no subjects will be taking neurally active or vasoactive medications. Any prior medications will be discontinued for at least 2 weeks.

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-02; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
To test whether 1 Liter volumes of intravenous or oral rehydration solution increase total blood volume and cardiac output, comparably improving the threshold for orthostatic intolerance | 1 week
  We will measure total blood volume, cardiorespiratory properties, plasma osmolarity and electrolytes before and after 1 hour after completing an intravenous infusion of normal saline. Hematocrit will be measure every 10 minutes for changes in blood volume. On a second day, we will measure total blood volume, cardiorespiratory properties, plasma osmolarity and electrolytes before and after 1 hour after ingesting 1 liter of oral rehydration solution. Hematocrit will be measure every 10 minutes for changes in blood volume.

CONTACTS AND LOCATIONS:
Overall Officials: Marvin S. Medow, Ph.D., Principal Investigator — New York Medical Collete
Locations (1):
- NewYork Medical College, Hawthorne, New York, United States

REFERENCES:
- See also: The Center for Hypotensioin — http://syncope.org